CLINICAL TRIAL: NCT04077398
Title: Volume Versus Concentration: a Prospective, Double Blind, Parallel Study to Compare the Clinical Effectiveness of Bilateral Quadratus Lumborum Blocks Using High Volume/Low Concentration or Low Volume/ High Concentration Local Anesthetic in Nephrectomies
Brief Title: Volume vs Concentration: Quadratus Lumborum Blocks With High Volume/Low Concentration or Low Volume/ High Concentration in Nephrectomies
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: covid interrupted initial start, then trainees involved finished program and no one took it on
Sponsor: Bruce Ben-David (Other)
Responsible Party: Sponsor-Investigator, Bruce Ben-David, Clinical Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY19070444
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Analgesia; Postoperative Pain; Block
MeSH Terms: conditions — Agnosia; Pain, Postoperative; Bites and Stings | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a prospective, randomized, double blinded, parallel trial at the University of Pittsburgh Medical Center (UPMC) Shadyside Hospital.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will be performed with software excel or spss. This randomization will be kept in an envelope. After the patient consents participation in the study, the investigator and the care provider will open the envelope and will perform the block according to the established in the randomization. The patient or the outcomes assessor will not have access to the volume and concentration used during the block. Will be the responsibility of investigators to keep in a safe place the information about the block received by the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- low volume High concentration group (Experimental): 1.Low Volume: 30 subjects randomized to Low Volume will receive bilateral Quadratus lumborum Block II. Each block of 0,75% ropivacaine x 15 mL + dexmedetomidine 0.4 mcg/kg (max dose 30 mcg for age <70, max dose 20 mcg for age >70) + dexamethasone 4 mg
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution
- high volume low concentration (Experimental): 2.High Volume: 30 subjects randomized to High Volume will receive bilateral Quadratus lumborum Block II. Each block of 0,375% ropivacaine x 30 mL + dexmedetomidine 0.4 mcg/kg (max dose 30 mcg for age <70, max dose 20 mcg for age >70) + dexamethasone 4 mg
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — There will be two groups, in order to compare two different sets of volumes with the same amount of drug. we will try to identify if it is better one volume over the other in terms of pain control and consume of opioids, as well the presence or absence of motor weakness.

SUMMARY:
The quadratus lumborum has since 2016 become standard of care for abdominal and retroperitoneal surgeries at UPMC-Shadyside Hospital, replacing paravertebral blocks, and as part of a broader multimodal analgesia institutional Enhanced Recovery After surgery protocol. Since the first description of this technique, several approaches to and anatomic targets within the quadratus lumborum plane have been described although their mechanism of action, spread, and relative clinical effectiveness remain areas of some debate. What is proposed here is to investigate the relative clinical effectiveness of the relationship high volume/low concentration of local anesthetic or low volume/ high concentration of local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-90 years old
2. Patients undergoing nephrectomy
3. Body Mass Index 19-36
4. Male and Female
5. All races
6. American Society of Anesthesiologist scale I, II, III

Exclusion Criteria:

1. Patient refusal
2. Pregnancy
3. Non-English speaking or inability to participate in the study
4. Patients with coagulopathy or With International Normalized Ratio >1,5 the day of the surgery.
5. Chronic steroid use
6. Chronic pain
7. Chronic opiate use

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
pain control over the next 72 hours after surgery: Visual analogue scale | 72 hours
  Visual analogue scale (0-10) measurement

SECONDARY OUTCOMES:
opioid consumption during the first 72 hours | 72 hours
  opioid consumption in morphine milliequivalents during the first 72 hours
time of the first opioid consumption after surgery | 24 hours
  time after surgery that patient takes to require opioid medication after surgery
100 feet walking | 48 hours
  time after surgery that the patient takes in order to be able to walk 100 feet
presence or absence of muscular weakness after Quadratus lumborum type 2 block | 24 hours
  muscular weakness is associated sometime with femoral quadratus muscle weakness

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC shadyside hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
there is no plan to share individual participant data.

REFERENCES:
- [Background] Murouchi T, Iwasaki S, Yamakage M. Quadratus Lumborum Block: Analgesic Effects and Chronological Ropivacaine Concentrations After Laparoscopic Surgery. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):146-50. doi: 10.1097/AAP.0000000000000349. PMID 26735154